CLINICAL TRIAL: NCT04633915
Title: A Comparison of Antibody Response Against SARS-CoV-2 in Hemodialysis and Non-dialysis Patients Diagnosed With COVID-19.
Brief Title: Antibody Response in Hemodialysis and Non-dialysis Patients Diagnosed With COVID-19.
Acronym: COV-HD
Status: Completed | Type: Observational
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Ekaterina Parshina, Principal investigator, MD, Saint Petersburg State University, Russia
Other Study IDs: COVID
Record Dates: First submitted 2020-11-15; First posted 2020-11-18 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Dialysis; Covid19
Keywords: antibodies; IgG; CKD; hemodialysis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for determination of antibodies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dialysis: Patients with CKD stage 5, treated with maintenance hemodialysis
- Healthy: Volunteers who are not dialysis-dependent

SUMMARY:
This is prospective cohort study aimed to compare antibody response against SARS-CoV-2 in dialysis patients and non-dialysis-dependent volunteers.

The research hypothesis is that dynamic of IgG antibodies against SARS-CoV-2 will differ in two groups.

To determine whether there is a statistically significant interaction between factors "group" and "time" on the titer of IgG antibodies against SARS-CoV-2, a two-way repeated measures ANOVA will be used.

DETAILED DESCRIPTION:
In both groups level of IgG antibodies against SARS-CoV-2 will be measured at the Day 1 (10 weeks from the date of first symptoms), Weeks 8 and 16 from the Day 1.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* SARS-CoV-2 infection within 10 weeks prior enrollment, confirmed by PCR or strongly suspected on computed tomography
* Providing informed consent

Exclusion Criteria:

* Refusal to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient ≥ 18 years old who were diagnosed with SARS-CoV-2 infection confirmed by PCR or strongly suspected on computed tomography within 10 weeks prior enrollment.
  Main group include patients with chronic kidney disease stage 5, receiving hemodialysis as a renal replacement therapy.
  The another group include volunteers who are not dialysis-dependent.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-07-18 (Actual)

PRIMARY OUTCOMES:
Anti-SARS-COV-2 IgG level | 16 weeks

SECONDARY OUTCOMES:
Proportion of people with detectable Anti-SARS-COV-2 IgG in study groups | Day 1, weeks 8, 16
Anti-SARS-COV-2 IgG level | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Petersburg State University Hospital, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided